CLINICAL TRIAL: NCT06362876
Title: The Effect of Breastfeeding Counseling Based on Motivational Interviewing Method in Women Having Cesarean Delivery
Brief Title: The Effect of Breastfeeding Counseling Based on Motivational Interviewing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Gozde Gokce Isbir, Professor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BAlis
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Breastfeeding Counseling Based on Motivational Interviewing
Keywords: Motivational Interviewing; Breastfeeding Consultancy; Breastfeeding; Midwife
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Breastfeeding Counseling Based on Motivational Interviewing (Experimental): Breastfeeding Counseling Based on Motivational Interviewing: An announcement was made on social media. Women who were willing to participate in the research and met the inclusion criteria were informed about the research and an appointment was made with them and they were scheduled to log in. All sessions were held with women individually and through online platforms. Motivational Interview-Based Breastfeeding Training Hypnobreastfeeding training program consists of 6 sessions and 4 parts. A total of 6 sessions were held with each woman, 3 implementation and 3 follow-ups.
  Interventions: Behavioral: Breastfeeding Counseling Based on Motivational Interviewing
- Standard Breastfeeding Consultancy (Experimental): Standard Breastfeeding Consultancy: The standard breastfeeding counseling program was prepared by the researchers with reference to the Breastfeeding Counseling Handbook published by the Ministry of Health of the Republic of Turkey in 2015. Training program consists of 6 sessions and 4 parts. A total of 6 sessions were held with each woman, 3 implementation and 3 follow-ups.
  Interventions: Behavioral: Standard Breastfeeding Consultancy

INTERVENTIONS:
Behavioral: Breastfeeding Counseling Based on Motivational Interviewing — Breastfeeding Counseling Based on Motivational Interviewing Program The breastfeeding counseling based on motivational interviewing program consists of 6 sessions and 4 hours. It includes information about breastfeeding, motivational preparation for the breastfeeding experience.
  Arms: Breastfeeding Counseling Based on Motivational Interviewing
Behavioral: Standard Breastfeeding Consultancy — Standart Breastfeeding Consultancy The standard breastfeeding consultancy program consists of 6session and 4 hours. It contains only information and applications about breastfeeding
  Arms: Standard Breastfeeding Consultancy

SUMMARY:
This research was planned to determine the effect of breastfeeding counseling based on motivational interviewing method and standard breastfeeding counseling on breastfeeding self-efficacy and breastfeeding results in women who had a cesarean section.

DETAILED DESCRIPTION:
This study was conducted between September 2023 and August 2024 as a single-blind randomized controlled study to determine the effect of breastfeeding counseling based on the motivational interview method and standard breastfeeding counseling on breastfeeding self-efficacy and breastfeeding results in women who had a cesarean section in Turkey. Participants who met the inclusion criteria were informed about the subject. The purpose of the study was explained to participants, and informed consent was obtained from all individuals who received motivational interviewing-based training or standard breastfeeding training. Data; When the research was approved, it was collected before the first counseling, in the first 48 hours after birth, and on the 14th day, 1st month and 3rd month after birth. CONSORT directive was followed in research planning

ELIGIBILITY:
Inclusion Criteria:

* Between September 2023 and August 2024
* Living in Turkey
* Seeing the poster about the research on social media and applying for the research
* Those between the ages of 18-40,
* Native speaker of Turkish,
* 34-40 weeks of pregnancy. between weeks,
* First pregnancy,
* Having a singleton pregnancy,
* Determining the type of birth as planned cesarean section,
* Do not have any chronic disease or pregnancy complications,
* There is no obstacle to breastfeeding,
* Does not have any psychiatric disease,
* Not receiving any individual, special training or counseling other than standard training and counseling regarding breastfeeding during pregnancy,
* Women who are ambivalent about breastfeeding

Exclusion Criteria:

* Not attending at least one of the counseling sessions to be held,
* Under 34 weeks and over 40 weeks,
* Participating in another training or receiving counseling regarding breastfeeding,
* Those who have health problems during the education process,
* Mother or baby has a health problem that will affect breastfeeding processes in the postpartum period,
* Those who have situations that may interrupt breastfeeding (hospitalization, medication use, separation from the baby, etc.),
* Leaving messages unanswered during the research process, not answering phone calls at least 5 times a week, and not returning to the researcher,
* Women who developed a psychological condition or psychiatric disorder during the research process

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Level of breastfeeding self-efficacy | 34-40 weeks of pregnancy
  Women's breastfeeding self-efficacy during pregnancy were evaluated with the Breastfeeding Self-efficacy Scale.
  This scale was developed by Dennis et al for fear after childbirth. The Turkish validity and reliability of the scale were performed by Tokat et al.This scale consisting of 14 items is a 5 point Likert type. The positive-meaning items are scored in reverse order. Therefore, the scores ranged from 14 to 70. The scale has no cutoff score, and high scores indicated higher breastfeedin self- efficacy.
  There are two versions of the scale used during pregnancy and postpartum. In both versions, the items are the same and the tenses change. In order to evaluate the Turkish validity and reliability of both antenatal and postnatal versions of the scale, language, structure and predictive validity analyzes were performed and the Cronbach's alpha value was found to be 0.87 for the antenatal measurement tool and 0.86 for the postnatal measurement tool.
Level of breastfeeding self-efficacy | Postpartum 24-48 hours
  Women's breastfeeding self-efficacy at the postpartum period were evaluated with the Breastfeeding Self-efficacy Scale.
  This scale was developed by Dennis et al for fear after childbirth. The Turkish validity and reliability of the scale were performed by Tokat et al. This scale consisting of 14 items is a 5 point Likert type. The positive-meaning items are scored in reverse order. Therefore, the scores ranged from 14 to 70. The scale has no cutoff score, and high scores indicated higher breastfeedin self- efficacy.
  There are two versions of the scale used during pregnancy and postpartum. In both versions, the items are the same and the tenses change. In order to evaluate the Turkish validity and reliability of both antenatal and postnatal versions of the scale, language, structure and predictive validity analyzes were performed and the Cronbach's alpha value was found to be 0.87 for the antenatal measurement tool and 0.86 for the postnatal measurement tool.
Level of breastfeeding self-efficacy | Postpartum 14. days
  Women's breastfeeding self-efficacy at the postpartum period were evaluated with the Breastfeeding Self-efficacy Scale.
  This scale was developed by Dennis et al for fear after childbirth. The Turkish validity and reliability of the scale were performed by Tokat et al. This scale consisting of 14 items is a 5 point Likert type. The positive-meaning items are scored in reverse order. Therefore, the scores ranged from 14 to 70. The scale has no cutoff score, and high scores indicated higher breastfeedin self- efficacy.
  There are two versions of the scale used during pregnancy and postpartum. In both versions, the items are the same and the tenses change. In order to evaluate the Turkish validity and reliability of both antenatal and postnatal versions of the scale, language, structure and predictive validity analyzes were performed and the Cronbach's alpha value was found to be 0.87 for the antenatal measurement tool and 0.86 for the postnatal measurement tool.
Level of breastfeeding self-efficacy | Postpartum 1. month
  Women's breastfeeding self-efficacy at the postpartum period were evaluated with the Breastfeeding Self-efficacy Scale.
  This scale was developed by Dennis et al for fear after childbirth. The Turkish validity and reliability of the scale were performed by Tokat et al. This scale consisting of 14 items is a 5 point Likert type. The positive-meaning items are scored in reverse order. Therefore, the scores ranged from 14 to 70. The scale has no cutoff score, and high scores indicated higher breastfeedin self- efficacy.
  There are two versions of the scale used during pregnancy and postpartum. In both versions, the items are the same and the tenses change. In order to evaluate the Turkish validity and reliability of both antenatal and postnatal versions of the scale, language, structure and predictive validity analyzes were performed and the Cronbach's alpha value was found to be 0.87 for the antenatal measurement tool and 0.86 for the postnatal measurement tool.
Level of breastfeeding self-efficacy | Postpartum 3. month
  Women's breastfeeding self-efficacy at the postpartum period were evaluated with the Breastfeeding Self-efficacy Scale.
  This scale was developed by Dennis et al for fear after childbirth. The Turkish validity and reliability of the scale were performed by Tokat et al. This scale consisting of 14 items is a 5 point Likert type. The positive-meaning items are scored in reverse order. Therefore, the scores ranged from 14 to 70. The scale has no cutoff score, and high scores indicated higher breastfeedin self- efficacy.
  There are two versions of the scale used during pregnancy and postpartum. In both versions, the items are the same and the tenses change. In order to evaluate the Turkish validity and reliability of both antenatal and postnatal versions of the scale, language, structure and predictive validity analyzes were performed and the Cronbach's alpha value was found to be 0.87 for the antenatal measurement tool and 0.86 for the postnatal measurement tool.
Breastfeeding Results Evaluation Form | Postpartum 24-48 hours
  The breastfeeding process evaluation form was created by researchers as a result of a literature review. The breastfeeding results evaluation form consists of 13 questions. It is a measurement tool that primarily determines individuals' current breastfeeding status, breastfeeding intentions in the first 6 months, breastfeeding confidence-sufficiency and breastfeeding importance scores. Breastfeeding confidence-sufficiency and breastfeeding importance scores are in the range of 0-10, and it is accepted that the higher the score, the higher the importance and value given.
Breastfeeding Results Evaluation Form | Postpartum 14. days
  The breastfeeding process evaluation form was created by researchers as a result of a literature review. The breastfeeding results evaluation form consists of 13 questions. It is a measurement tool that primarily determines individuals' current breastfeeding status, breastfeeding intentions in the first 6 months, breastfeeding confidence-sufficiency and breastfeeding importance scores. Breastfeeding confidence-sufficiency and breastfeeding importance scores are in the range of 0-10, and it is accepted that the higher the score, the higher the importance and value given.
Breastfeeding Results Evaluation Form | Postpartum 1. month
  The breastfeeding process evaluation form was created by researchers as a result of a literature review. The breastfeeding results evaluation form consists of 13 questions. It is a measurement tool that primarily determines individuals' current breastfeeding status, breastfeeding intentions in the first 6 months, breastfeeding confidence-sufficiency and breastfeeding importance scores. Breastfeeding confidence-sufficiency and breastfeeding importance scores are in the range of 0-10, and it is accepted that the higher the score, the higher the importance and value given.
Breastfeeding Results Evaluation Form | Postpartum 3. month
  The breastfeeding process evaluation form was created by researchers as a result of a literature review. The breastfeeding results evaluation form consists of 13 questions. It is a measurement tool that primarily determines individuals' current breastfeeding status, breastfeeding intentions in the first 6 months, breastfeeding confidence-sufficiency and breastfeeding importance scores. Breastfeeding confidence-sufficiency and breastfeeding importance scores are in the range of 0-10, and it is accepted that the higher the score, the higher the importance and value given.

CONTACTS AND LOCATIONS:
Overall Officials: Gozde Gokce Isbir, Professor, Principal Investigator — Mersin University
Locations (1):
- Mersin University, Mersin, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Breastfeeding Self-Efficacy Scale: Psychometric Assessment of the Short Form — https://doi.org/10.1177/0884217503258459
- See also: The Relation Between Breastfeeding Self-Efficacy and Breastfeeding Successes of Mothers — https://jer-nursing.org/jvi.aspx?pdir=jern&plng=eng&un=JERN-08208&look4=